CLINICAL TRIAL: NCT07338357
Title: A Single-Center Clinical Study Evaluating the Safety and Preliminary Efficacy of CLL-1 CAR-T in the Treatment of Children With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Clinical Study of CLL-1 CAR-T in the Treatment of Children With R/R AML
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Principal Investigator, Yunyan He, PhD, First Affiliated Hospital of Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG-CT-25-012
Record Dates: First submitted 2025-12-22; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: AML (Acute Myeloid Leukemia); CAR-T
Keywords: R/R AML; CAR-T
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T (Experimental): CAR-T therapy
  Interventions: Biological: CAR-T

INTERVENTIONS:
Biological: CAR-T — A infusion of CLL-1 CAR-T cells following a lymphodepleting chemotherapy regimen.

SUMMARY:
A study to evaluate the safety and preliminary efficacy of CLL-1-targeted CAR-T cell therapy in children aged 3 to 18 years with relapsed or refractory acute myeloid leukemia (r/r AML).

DETAILED DESCRIPTION:
It's a single-center, single-arm, investigator-initiated clinical study. After thorough consideration and signing of the informed consent form by the subject and/or their legal guardian(s), subjects meeting the eligibility criteria during the screening period will provide blood samples for CAR-T manufacturing. Following lymphodepleting chemotherapy, CAR-T cell infusion will be administered on D0.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the ICF and are expected to complete the study's follow-up examinations and procedures.
2. Aged 3 to 18 years (inclusive), and body weight ≥10 kg.
3. Diagnosis of AML according to the 2016 WHO classification, meeting the diagnostic criteria for relapse and refractoriness as per the "Chinese Guidelines for Diagnosis and Treatment of Relapsed/Refractory Acute Myeloid Leukemia (2017 Edition)", and currently having no clinically relevant treatment options or suitable registered clinical trials available.
4. Confirmation of CLL-1 expression ≥50% on AML blasts by flow cytometry.
5. Recovery from toxicities of prior therapies.
6. Karnofsky score (for age ≥16 years) ≥70 or Lansky score (for age <16 years) ≥50 at screening, and an expected survival >3 months.
7. Suitable function of the liver, kidneys, hematological system, lungs and heart is required.
8. Females subjects of childbearing potential must have a negative blood pregnancy test at screening and agree to use effective contraception during the study and within 1 year after the last dose of study drug.
9. Male subjects with reproductive potential must agree to use barrier contraception or practice complete abstinence until 1 year after the last study treatment.
10. Eligible blood cell specimen can be provided.

Exclusion Criteria:

1. Diagnosis of APL.
2. History of other malignancies within 3 years prior to screening, except for adequately treated carcinoma in situ of the cervix, papillary thyroid carcinoma, basal cell or squamous cell skin cancer, localized prostate cancer treated with radical surgery, and ductal carcinoma in situ treated with radical surgery.
3. Evidence of CNS involvement or cranial nerve pathology.
4. Subjects with active infections such as hepatitis B, hepatitis C, etc., are to be excluded.
5. Subjects with a history of severe allergies or known allergy to any drug component included in this study are to be excluded.
6. Subjects with severe cardiac diseases, refractory hypertension, active neurological autoimmune or inflammatory diseases, clinically significant active cerebrovascular disease, oncologic emergencies requiring urgent intervention, acute or chronic GVHD, or any uncontrolled infections requiring antibiotic therapy, etc., are unsuitable for enrollment.
7. Previous organ transplant or planned organ transplant (except for hematopoietic stem cell transplantation).
8. Received allo-HSCT within 6 weeks prior to screening.
9. Subjects who have recently undergone major surgery or plan to undergo major surgery, excluding diagnostic procedures and biopsies.
10. Subjects with severe mental disorders, alcoholism, or drug abuse.
11. Subjects who, in the judgment of the investigator, have other conditions that make them unsuitable for enrollment.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events | Up to 2 years.
  Proportion of subjects experiencing all kinds of treatment-related AEs.

SECONDARY OUTCOMES:
Overall Response Rate | Up to 2 years.
  Proportion of subjects achieving CR, CRi, morphologic leukemia-free state (MLFS), or PR.
Duration of Response | Up to 2 years.
  Time from first assessment of CR, CRi, MLFS, or PR to first assessment of disease recurrence/progression or death from any cause.
Relapse-Free Survival | Up to 2 years.
  For subjects achieving CR, CRi, or CR MRD-only. Time from achievement of response to relapse or death (any cause).
Event-Free Survival | Up to 2 years.
  For all subjects. Time from cell infusion to treatment failure, relapse, or death (any cause).
Overall Survival | Up to 2 years.
  For all subjects. Time from cell infusion to death from any cause.
Proportion of CLL-1-Positive Tumor Cells | Up to 2 years.
  Changes in the proportion of CLL-1-positive tumor cells after CLL-1 CAR-T infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Yunyan He, PhD, Principal Investigator — First Affiliated Hospital of Guangxi Medical University

IPD SHARING:
Plan to Share IPD: No